CLINICAL TRIAL: NCT04751786
Title: First-in-human Phase I Dose Escalation Study Assessing Safety, Tolerability and Preliminary Efficacy of Immunomodulatory Nanoparticles
Brief Title: Dose Escalation Study of Immunomodulatory Nanoparticles
Acronym: PRECIOUS-01
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: CATO-SMS (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NL 72876.091.20; 2017-002568-41 (EudraCT Number)
Record Dates: First submitted 2020-12-11; First posted 2021-02-12 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Advanced Solid Tumor
Keywords: Advanced solid tumor; No standard treatment available; Phase I dose escalation study; IHC-confirmed NY-ESO-1 positivity

STUDY DESIGN:
Intervention Model Description: Eligible subjects will receive three i.v. infusions of PRECIOUS-01 at a 3-weekly interval in three dose-finding cohorts (low: 0.4 mg/kg, intermediate: 0.8 mg/kg, and high: 1.6 mg/kg fixed doses). Subjects will be monitored for safety and the occurrence of Dose-Limiting Toxicities (DLTs). A 3+3 design is used for the dose escalation steps. Three subjects will be enrolled sequentially per cohort. If the maximum tolerated dose (MTD) is not reached in the planned dose escalation cohorts, the RP2D will be based on the observed safety and immune modulatory activity as pharmacodynamic parameter supporting the RP2D. The sample size is based on the determination of the MTD/RP2D. In order to collect sufficient information regarding changes in immune related parameters as readout for pharmacodynamics of the particles, it is planned to extend the two highest dosing cohorts to a total of six subjects or to extend the highest dosing cohort to a total of nine subjects, depending on observed toxicity.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- PRECIOUS-01 (Experimental): Eligible subjects will receive three i.v. infusions of PRECIOUS-01 at a 3-weekly interval in three dose-finding cohorts (low: 0.4 mg/kg, intermediate: 0.8 mg/kg, and high: 1.6 mg/kg fixed doses). Subjects will be monitored for safety and the occurrence of Dose-Limiting Toxicities (DLTs). A 3+3 design is used for the dose escalation steps. Three subjects will be enrolled sequentially per cohort. If the maximum tolerated dose (MTD) is not reached in the planned dose escalation cohorts, the RP2D will be based on the observed safety and immune modulatory activity as pharmacodynamic parameter supporting the RP2D. The sample size is based on the determination of the MTD/RP2D. In order to collect sufficient information regarding changes in immune related parameters as readout for pharmacodynamics of the particles, it is planned to extend the two highest dosing cohorts to a total of six subjects or to extend the highest dosing cohort to a total of nine subjects, depending on observed toxicity
  Interventions: Drug: PRECIOUS-01

INTERVENTIONS:
Drug: PRECIOUS-01 — Subjects will be enrolled in one of three dosing cohorts (three subjects per cohort for the planned dose escalation with a planned extension to a total of six subjects for the two highest dosing cohorts for the evaluation of the pharmacodynamic effects of PRECIOUS-01 for determination of the RP2D, if MTD is not reached).

SUMMARY:
PRECIOUS-01 is an immunomodulating agent composed of the invariant natural killer T cell (iNKT) activator threitolceramide-6 (ThrCer6, IMM60) and the New York Esophageal Squamous Cell Carcinoma-1 (NY-ESO-1) cancer-testis antigen peptides encapsulated in a poly(lactic-co-glycolic acid) (PLGA) nanoparticle.

PRECIOUS-01 is being developed for the treatment of patients with NY-ESO-1-positive cancers.

DETAILED DESCRIPTION:
In the rapidly evolving treatment landscape of advanced solid tumors, immunotherapeutic approaches have revolutionized cancer care for patients. Despite these advances, there is an undiminished need for the development of novel immunotherapeutic treatment modalities that are able to orchestrate effective anti-tumor immune responses. The investigators study a new class of immunomodulatory nanomedicines: PLGA nanoparticles loaded with a tumor antigen and an iNKT cell agonist.

PLGA is a biodegradable polymer with minimal (systemic) toxicity, approved by the Food and Drug Administration (FDA) as well as the European Medicines Agency (EMA) to be used in various drug-carrying platforms.Tumor antigens and immunomodulatory molecules can be co-encapsulated in PLGA-based nanoparticles. In preclinical studies, these PLGA-based nanoparticles can induce anti-tumor immune responses. The investigators aim to explore PLGA-based nanoparticles containing the tumor antigen NY-ESO-1 and the iNKT cell activator IMM60 for their capacity to induce anti-tumor responses in cancer patients.

NY-ESO-1 is a cancer-testis antigen normally expressed in testicular germ cells and trophoblasts of the placenta. However, NY-ESO-1 is also expressed in a wide range of cancers with a high incidence (around 25-30% of several [advanced] cancers, such as melanoma [40%], lung [2-32%], bladder [32-35%], and ovarian [30%] cancer). NY-ESO-1 is able to elicit immune responses. Patients who have NY-ESO-1-positive tumors have spontaneous or vaccine-induced humoral and cellular immune responses against this antigen. Therefore, NY-ESO-1 is considered to be a suitable tumor antigen for further clinical evaluation. Clinical trials have already shown the safety and tolerability of the NY-ESO-1 protein and peptides in patients with advanced cancer.

In order to generate NY-ESO-1-directed immune responses, the NY-ESO-1 protein is taken up by antigen-presenting cells (APCs) and processed in small protein fragments, peptides. Particular peptides can bind to patient-specific HLA molecules and, subsequently, this HLA-peptide complex is recognized at the cell membrane by the T cell receptor (TCR) of T cells. Once the TCR specifically binds to the HLA-peptide complex, the T cell becomes stimulated and exerts its function, i.e. tumor cell killing by CD8+ T cells. In 1, an overview of the peptides known to bind to certain HLA alleles and recognized by T cells, either by CD4+ or by CD8+ T cells, is presented.

Particulate vaccines are known to elicit better immune responses due to higher uptake by APCs. Encapsulating antigens and adjuvants within the same polymeric nanoparticle can enhance T cell responses. In earlier studies, the NY-ESO-1 whole protein was encapsulated in adjuvant ISCOMATRIX and shown to induce specific T cell responses in a majority of patients. iNKT cell agonists are more suitable adjuvants due to their higher activity in low doses and activation of DCs by iNKT cells. In this respect, the investigators will employ PLGA nanoparticles loaded with the NY-ESO-1 antigen and the iNKT cell agonist IMM60 as a co-delivery system.

To facilitate NY-ESO-1 antigen encapsulation, long (85-111(peptide #2) and 117-143(peptide #3)) and short (157-165(peptide #4)) peptides will be incorporated into nanoparticles. In combination, the three selected NY-ESO-1-derived peptides are presented in 80% of the class I and class II HLA alleles of the European population. Similar peptides (79-116 and 118-143) were previously loaded onto DCs together with α-GalCer and delivered to cancer patients in a recent clinical trial. The results of that trial demonstrated iNKT cell expansion, CD4+ T cell responses against the 118-143 peptide in 7/8 patients, and CD8+ T cell responses against the 79-116 peptide in 3/8 patients (Gasser, Sharples et al. 2018). Here, an additional short peptide (157-165) is included, which is presented by the highly prevalent HLA-A2.1 molecule. Hence, higher CD8+ T cell responses against this epitope and superior activation of human iNKT cells by IMM60 are expected due to co-encapsulation.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older at time of signing informed consent.
2. Performance status (ECOG 0 or 1).
3. Estimated life expectancy of at least 6 months.
4. Histologically or cytologically confirmed advanced and /or metastatic solid tumor with progressive disease at baseline, for whom no standard treatment is available.
5. IHC-confirmed NY-ESO-1 positivity prior to screening (cut-off value: 1% positive cells) on (archival) tumor tissue, per local laboratory guidelines.
6. Subject with evaluable disease per RECIST v1.1.
7. Adequate hematologic, renal and liver function as defined by laboratory values performed within 14 days of start of treatment:

   1. Hemoglobin (Hb) ≥ 6 mmol/L;
   2. Absolute Lymphocyte Count (ALC) > 0.8 x 109/L;
   3. Absolute Neutrophil Count (ANC) ≥ 1.5 × 109/L;
   4. Platelet count > 100 x 109/L;
   5. Creatinine level within normal institutional limit;
   6. Serum bilirubin < 25 μmol/L;
   7. Serum Lactic Acid Dehydrogenase (LDH) ≤ Upper Limit of Normal range (ULN);
   8. Alkaline Phosphatase (ALP), Aspartate Aminotransferase (AST), and Alanine Aminotransferase (ALT) ≤ ULN unless related to liver metastasis (in which case levels should be < 3 ULN).
8. Previous therapy-derived toxicities should be resolved to Grade < 2 according to CTCAE v5.0, with exceptions for alopecia.
9. All subjects of childbearing potential (defined as < 2 years after last menstruation or not surgically sterile) must have a negative highly sensitive pregnancy test at screening (urine/serum) and agree to use a highly effective method for contraception according to the EU Clinical Trial Facilitation Group guidance from time of signing the informed consent form (ICF) until at least 120 days after the last administration of PRECIOUS-01. The partners of subjects with childbearing potential must also apply contraceptive methods, and are recommended not to donate sperm.
10. Before registration, ability of subject to give written informed consent according to International Council for Harmonisation (ICH) Good Clinical Practice (GCP), and national rules/local regulations.
11. Expected adequacy of follow-up.

Exclusion Criteria:

1. Second malignancy in the previous 2 years, with the exception of adequately treated in situ carcinoma of the cervix uteri and basal or squamous cell carcinoma of the skin,
2. Clinical suspicion or radiological evidence of active brain metastases. Patients with brain metastases that have been treated previously and are proven stable (computed tomography [CT] or magnetic resonance imaging [MRI] < 30 days) and without steroids for > 3 months are allowed.
3. Subjects with thromboembolic events within the past year.
4. Subjects on any other anticancer therapy (cytotoxic, biologic or investigational agents), unless at least 4 weeks (or 5 half-lives, whichever is shorter, 6 weeks for mitomycin-C or nitrosoureas), have elapsed since the last dose before the first administration of PRECIOUS-01. At least 4 weeks should have elapsed since receiving palliative radiotherapy. Chronic treatment with non-investigational gonadotropin-releasing hormone analogs or other hormonal or supportive care is permitted.
5. Subjects with major surgery within 4 weeks before initiating treatment or with minor surgical procedure within 7 days before initiating treatment (except for port-a-cath or central line i.v. placement, or biopsy), or anticipation of the need for major surgery during the course of the trial treatment.
6. Concomitant use of oral or i.v. immunosuppressive drugs. Inhaled, topical or intranasal steroids and adrenal replacement steroids < 10 mg/day (prednisone equivalent) are permitted in the absence of auto-immune disease.
7. Uncontrolled infectious disease, i.e. negative testing for human immunodeficiency virus (HIV), Hepatitis B Virus (HBV), Hepatitis C Virus (HCV) and syphilis (Treponema Pallidum Hemagglutination Assay [TPHA]).
8. (Systemic) autoimmune disease such as, but not limited to, inflammatory bowel disease, multiple sclerosis and lupus. Subjects with type 1 diabetes mellitus, hypothyroidism after autoimmune thyroiditis and skin disorders (eczema and psoriasis) are not excluded.
9. History of clinically significant cardiovascular disease (≤ 6 months prior to Day 1 on trial) such as stroke, Transient Ischemic Attack (TIA), unstable angina, New York Heart Association (NYHA) Grade II or greater congestive heart failure, myocardial infarction, uncontrolled hypertension, cardiac arrhythmia requiring medication, relevant pathological ECG findings or uncontrolled hypertension (systolic > 150 mm Hg and/or diastolic > 100 mm Hg).
10. Serious (bleeding and clotting) condition(s) that may interfere with safe administration of PRECIOUS-01.
11. Abnormal or clinically significant coagulation parameters at the discretion of the Clinical Investigator, i.e.:

    1. Prothrombin Time - International Normalized Ratio (PT-INR)
    2. Activated Partial Thromboplastin Time (APTT)
    3. Subjects being treated with anticoagulants are excluded if the coagulation parameters are outside the therapeutic intervals as described in the Summary of Product Characteristics (SmPC) for the administered treatment.
12. Evidence of any other conditions (such as psychological/familial sociological/geographical issues, psychiatric illness, infectious diseases, physical examination or laboratory findings) that may interfere with the planned treatment, affect subject compliance or place the subject at high risk from treatment-related complications. These conditions must be discussed with the subject before registration in the trial.
13. History of severe allergic episodes and/or Quincke's edema.
14. Prior allogeneic tissue/solid organ transplant, stem cell or bone marrow transplant.
15. Known hypersensitivity to any component of PRECIOUS-01.
16. Pregnant or lactating women. A serum pregnancy test should be performed within 7 days prior to start of trial treatment for confirmation in case of childbearing potential.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2021-01-11 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Safety of PRECIOUS-01 | From enrollment up to and including 21 days after last PRECIOUS-01 administration (all AEs). Related AEs and SAEs will be followed up until 17 weeks after end of treatment.
  The incidence of treatment-emerging Adverse Events (AEs) according to the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) v5.0 reporting severity and relatedness
Multiplex immunohistochemistry assay to gain insight into the composition of immune cell subsets | At baseline and at the end of Cycle 3 (each cycle is 21 days)
  To analyze the immunological composition in tumor biopsies using an established immunohistochemistry (IHC) assay for the detection of CD3, CD8, FoxP3, CD45RO and CD20 positive cells; these results will support the decision on the RP2D as part of the planned trial.

SECONDARY OUTCOMES:
Recommended Phase 2 Dose (RP2D) | From enrollment up to and including 21 days after last PRECIOUS-01 administration. Side effects will be followed up until 17 weeks after end of treatment.
  To determine the Recommended Phase 2 Dose (RP2D) of PRECIOUS-01 for a subsequent Phase II trial.
Immunological responses in blood | From study initiation up to and including the database lock, which is estimated to be 24 months later
  Occurrence and magnitude of functional responses of iNKT cells and T cells will be studied. Serum cytokine levels will be determined by cytokine bead array. T cell specificity will be tested by multimer analysis. DC, iNKT cell, and NK cell activation status and functionality studies (cytokine responses) by flowcytometry. PAXgene blood will be collected before and 24 hours after every IMP administration. mRNA levels for IFN-related genes will be determined by qPCR. Anti-NY-ESO-1 antibodies will be studied.

OTHER OUTCOMES:
Best Overall Response | From study initiation up to and including the database lock, which is estimated to be 24 months later
  Response Evaluation Criteria in Solid Tumors (RECIST) v1.1. is used to evaluate the best overall response.

CONTACTS AND LOCATIONS:
Overall Officials: Petronella B. Ottevanger, MD, PhD, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboudumc, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will be listed by measure and time point.
Supporting Information: Study Protocol, SAP

REFERENCES:
- [Background] Dolen Y, Kreutz M, Gileadi U, Tel J, Vasaturo A, van Dinther EA, van Hout-Kuijer MA, Cerundolo V, Figdor CG. Co-delivery of PLGA encapsulated invariant NKT cell agonist with antigenic protein induce strong T cell-mediated antitumor immune responses. Oncoimmunology. 2015 Aug 12;5(1):e1068493. doi: 10.1080/2162402X.2015.1068493. eCollection 2016. PMID 26942088
- [Derived] Creemers JHA, Pawlitzky I, Grosios K, Gileadi U, Middleton MR, Gerritsen WR, Mehra N, Rivoltini L, Walters I, Figdor CG, Ottevanger PB, de Vries IJM. Assessing the safety, tolerability and efficacy of PLGA-based immunomodulatory nanoparticles in patients with advanced NY-ESO-1-positive cancers: a first-in-human phase I open-label dose-escalation study protocol. BMJ Open. 2021 Nov 30;11(11):e050725. doi: 10.1136/bmjopen-2021-050725. PMID 34848513